CLINICAL TRIAL: NCT04874714
Title: Prospective, Randomized, Placebo-controlled, Multi-center Trial Comparing the Efficacy and Safety of Subcutaneous Immunotherapy With a Mixture of Grasses and Mites at Adequate Doses Versus Monotherapy, for the Treatment of Allergy
Brief Title: Efficacy and Safety Evaluation for the Treatment of Asthma and Allergic Rhinitis/Rhinoconjunctivitis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to the low recruitment rate since the start of the trial
Sponsor: Inmunotek S.L. (Industry)
Collaborators: BioClever 2005 S.L. (Other); NTS hub S.L (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DMV01-SIT-015; 2018-003715-22 (EudraCT Number)
Record Dates: First submitted 2021-03-26; First posted 2021-05-06 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Allergic Rhinoconjunctivitis; Perennial Allergic Rhinitis; House Dust Mite Allergy; Pollen Allergy
Keywords: Rhinitis/ Rhinoconjunctivitis; Mild to moderate asthma; Allergy; Immunotherapy; Mite; Pollen; Vaccine
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Dust Mite Allergy; Rhinitis, Allergic, Seasonal; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, placebo-controlled, multi-center trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: During the trial, both the investigator and the included subjects will be unaware of the treatment each subject is receiving.
  The person in charge of data analysis will also not know the treatment assigned to each subject until the database has been closed.
  So that neither the subject nor the investigator knows what treatment each subject is receiving, all the trial medication is identical in terms of outer packaging and appearance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MM09-MG01(30.000-30.000) (Experimental): 30,000 AU/mL of MM09 and 30,000 AU/mL of MG01 of subcutaneous immunotherapy once a month for 11 months
  Interventions: Biological: MM09-MG01(30.000-30.000)
- MG01(30.000) (Experimental): 30,000 AU/mL of MG01 of subcutaneous immunotherapy once a month for 11 months
  Interventions: Biological: MG01(30.000)
- MM09(30.000) (Experimental): 30,000 AU/mL of MM09 of subcutaneous immunotherapy once a month for 11 months
  Interventions: Biological: MM09(30.000)
- Placebo subcutaneous (Placebo Comparator): The same solution, presentation, method of administration, frequency, and duration as the active treatment, but without active ingredients.
  Interventions: Biological: Placebo subcutaneous

INTERVENTIONS:
Biological: MM09-MG01(30.000-30.000) — Mite mixture (Dermatophagoides pteronyssinus and Dermatophagoides farinae) with a concentration of 30,000 AU / mL and grasses mixture (Phleum pratense, Holcus lanatus, Poa pratensis, Festuca elatior, Lolium perenne and Dactylis glomerata) with a concentration of 30,000 AU / mL: Purified allergenic extract, adsorbed in aluminum hydroxide and polymerized with glutaraldehyde
  Arms: MM09-MG01(30.000-30.000)
Biological: MG01(30.000) — Grasses mixture (Phleum pratense, Holcus lanatus, Poa pratensis, Festuca elatior, Lolium perenne and Dactylis glomerata) with a concentration of 30,000 AU / mL: Purified allergenic extract, adsorbed in aluminum hydroxide and polymerized with glutaraldehyde
  Arms: MG01(30.000)
Biological: MM09(30.000) — Mite mixture (Dermatophagoides pteronyssinus and Dermatophagoides farinae) with a concentration of 30,000 AU / mL: Purified allergenic extract, adsorbed in aluminum hydroxide and polymerized with glutaraldehyde
  Arms: MM09(30.000)
Biological: Placebo subcutaneous — The same solution, presentation, method of administration, frequency, and duration as the active treatment, but without active ingredients.
  Arms: Placebo subcutaneous

SUMMARY:
Prospective, randomized, placebo-controlled, multicenter of 3 active treatment groups, compared to 1 placebo group, for the determination of the efficacy and safety of subcutaneous immunotherapy in patients with mild to moderate asthma and allergic rhinitis/rhinoconjunctivitis (intermittent or persistent) due to hypersensitivity to house dust mites (Dermatophagoides pteronyssinus and / or D. farinae) and grass pollen

DETAILED DESCRIPTION:
Double blind, parallel placebo-controlled study. The subjects will receive medication during 11 months

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have signed the informed consent
2. Subjects with a confirmed medical history of asthma (intermittent or persistent mild-moderate, controlled), as defined by GEMA 5 with moderate-severe rhinitis / rhinoconjunctivitis (intermittent or persistent) according to the ARIA classification caused by polysensitization to grass pollen and mites (D. pteronyssinus and / or D. farinae). The diagnosis of asthma will be valid from 24 months prior to signing the informed consent.
3. Subjects with a positive prick test (major diameter of the papule ≥ to 5 mm) to a standardized extract of grass pollen mixture, or to one of the components of the mixture (Dactilys glomerata, Poa pratensis, Holcus lanatus, Festuca elatior, Phleum pratense and Lolium perenne) and to an extract of D. pteronyssinus and / or D. farinae. Results will be valid 12 months prior to signing the informed consent.
4. Specific IgE (CAP or Immulite) against one of the components of the mixture of grasses, preferably Phleum pratense or a mixture of grasses and mites (D. pteronyssinus and / or D. farinae) or one or more of the molecular components of allergenic sources with a value > 3,5 KU / L. Results will be valid 12 months prior to signing the informed consent.
5. Subjects will preferably be sensitive to study allergens (Dermatophagoides and grasses). In the case of subjects sensitized to other aeroallergens, only those with the following characteristics (results valid up to 12 months prior to signing of the informed consent) can be included in the study:

   1. Subjects with a positive prick test for Blomia tropicalis and Lepidoglyphus destructor, whose maximum values of specific IgE are 3.5 KU/L and do not exceed or equal the values of the allergens of the study (Dermatophagoides and grasses).
   2. Subjects with a negative prick test to epithelium, whose specific IgE values are < 0.35 KU/L. Subjects with occasional exposure and symptomatology to epithelium may be included with a positive prick test regardless of the value of the specific IgE.
   3. Subjects with a positive prick test for non-coestational pollens, whose maximum values of specific IgE are 17.5 KU / L and do not exceed or equal the values of the allergens of the study (Dermathophagoids and grasses) and who also do not present exacerbations in the pollen season.
6. Subjects with a negative prick test for fungi. If the specific IgE determination has been made, the result shall be < 0,35 KU/L.
7. Subjects with a negative prick test for coestacional pollens with grasses. If the specific IgE determination has been made, the result shall be < 0,35 KU/L.
8. Subjects aged between 12 and 65 years, inclusive.
9. Subjects capable of complying with the dosing regimen.
10. Women of childbearing age (from menarche) should submit a urine pregnancy test with a negative result at the time of enrolment in the trial.
11. Women of childbearing potential should commit to using an adequate method of contraception. Medically acceptable methods of contraception are intrauterine devices placed at least 3 months in advance, surgical sterilization (for example, tubal ligation), barrier methods, or the use of oral contraceptives.
12. Subjects who have a smartphone to record symptoms and medication.

Exclusion Criteria:

1. Subjects who have received prior immunotherapy treatment in the preceding 5 years for any aeroallergen.
2. Patients in whom immunotherapy may be the object of an absolute general contraindication according to the criteria of the Immunotherapy Committee of the Spanish Society of Allergy and Clinical Immunology and the European Allergy and Clinical Immunology Immunotherapy Subcommittee cannot be included.
3. Subjects with severe or uncontrolled asthma, and / or with a FEV1 <70% with respect to the reference value despite adequate pharmacological treatment at the time of inclusion in the trial.
4. Subjects who have previously presented a serious secondary reaction during the performance of diagnostic skin tests using the prick test.
5. Subjects under treatment with ß-blockers.
6. Subjects under treatment with immunosuppressive or biological drugs.
7. Clinically unstable subjects at the time of inclusion in the trial (respiratory infection, feverish process, acute urticaria, etc.).
8. Subjects with chronic urticaria in the past 2 years, severe anaphylaxis, or a history of hereditary angioedema.
9. Subjects who have any pathology in which the administration of adrenaline is contraindicated (hyperthyroidism, HT, heart disease, etc.).
10. Subjects with some other disease not related to moderate rhinoconjunctivitis or asthma, but of potential severity and that may interfere with treatment and follow-up (epilepsy, psychomotor disorder, diabetes, malformations, subjects who underwent multiple surgeries, kidney disease...), according to investigator's criteria.
11. Subjects with autoimmune disease (thyroiditis, lupus, etc.), tumour diseases or with a diagnosis of immunodeficiencies.
12. Subject whose condition prevents him / her from offering cooperation and or who resents severe psychiatric disorders, according to investigator criteria.
13. Subjects with known allergies to other investigational product components other than grass pollen or mites.
14. Subjects with diseases of the lower respiratory tract other than asthma such as emphysema or bronchiectasis.
15. Pregnant or lactating women.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2023-10-09 (Actual); Study Completion 2023-10-09 (Actual)

PRIMARY OUTCOMES:
CSMS: Combined Symptoms and Medication Score | 12 months
  Evaluation of the number of symptoms and the consumption of medication necessary for the control of such symptoms in asthma and rhinitis / rhinoconjunctivitis of each subject during the trial, of the groups with each other and with respect to placebo.
  - The endpoint for each asthma and rhinitis / rhinoconjunctivitis symptom will be as follows: 0 = No symptoms; 1 = Mild; 2 = Moderate; 3 = Severe
  Total daily symptom score = 0-3
  * The asthma medication will be scored based on the therapeutic step in which drugs are included in the GEMA 5 guide.
  * The rhinitis / rhinoconjunctivitis medication score: 0 = No medication; 1 = oral or topical (eyes or nose) non-sedative H1 antihistamines (H1A); 2 = intranasal corticosteroids (INS) with / without H1A; 3 = oral corticosteroids with/without (INS), with/without H1A
  Total daily medication score = 0-3

SECONDARY OUTCOMES:
Medication-free days | 12 months
  Number of days that the subjects need no medication
Symptom-free days | 12 months
  Number of days that the subjects have no symptom
Respiratory function_FEV1 | 12 months
  Measurement of Forced Expiratory Volume in 1 Second (FEV1) %
Respiratory function_PEF | 12 months
  Peak Expiratory Flow (PEF) [velocity]
Asthmatic exacerbations | 12 months
  Time elapsed until the first appearance of asthmatic exacerbations, number, duration and severity.
Immunological parameters | 12 months
  Analyses of total and specific IgE, specific IgE index / total IgE and specific IgG4
Visual Analogue Scale (VAS) | 12 months
  Visual Analogue Scale in which the subject has to indicate in a straight line of 10cm how he/she feels regarding to his allergy symptoms. Being left side (0) = very bad and right side (10) = very well
Quality of life associated with rhinitis | 12 months
  The quality of life associated with rhinitis will be measured following the test ESPRINT-15.
  The scoring of the questionnaire will be carried out as follows: The global sum of the scores (ranging from "0 = nothing has bothered me" to "6 = it has bothered me a lot") of the 14 items plus the score given in the general questionnaire (ranging from "0 = Excellent" to "4 = Bad"). This sum is divided by the total number of items (15 items).
  The interpretation of the scores is between 0 (low impact) and 6 (high impact).
Quality of life associated with asthma | 12 months
  The quality of life associated with asthma will be measured following the ACQ questionnaire.
  The ACQ questionnaire consists of 7 questions (ACQ-7) or 6 questions (ACQ-6). In questions 1-6, patients recall their experience during the last 7 days and answer using a scale of 7 points (from 0 = fully controlled to 6 = extremely poorly controlled). The seventh question, which refers to the% FEV1 of the reference value, must be completed by an employee of the site. The questionnaire score is the mean of the 7 responses (ACQ-7) or 6 responses (ACQ-6).
  The interpretation of the scores is as follows:
  * Less than or equal to 0.75: Adequate control of asthma
  * From 0.75 to 1.50: Partially controlled asthma
  * More than 1.50: Inadequate asthma control
Consumption of health resources | 12 months
  For each patient, the number of times that due to allergy symptoms has done the following will be counted:
  * have visited the family doctor
  * have made an unscheduled visit to the specialist
  * has gone to the emergency room
  * has been hospitalized
  * have needed to contact the doctor by phone
Security parameters | 12 months
  Global rate and severity of AE per administration and per subject
Number of Local Adverse Reactions | 12 months
  Local adverse reactions are those that appear at the site of the administration. They are classified into: Inmediate (it appears during the first 30 minutes from the administration of investigational product) and Late (it appears after the first 30 minutes from the administration of investigational product)
  Local adverse reactions are considered if a papule > 5 cm in diameter occurs in the first 30 minutes after administration (immediate local reactions) or > 10 cm if it is later (late local reactions).
Number of Systemic Adverse Reactions | 12 months
  Systemic adverse reactions are those that appear in other parts of the body other than the site of administration.Their severity will be classified following the indications proposed by the World Allergy Organization (WAO) in 2010, measured according to the following grades:
  * Grade 0: Absence of symptoms or nonspecific symptoms.
  * Grade 1: Signs or symptoms present in a system / organ (cutaneous, Upper respiratory tract, Conjunctival or Other)
  * Grade 2: Signs and symptoms of 2 or more organs / systems listed in Grade 1, or; Lower airway disease, or; Gastrointestinal symptoms, or; Other
  * Grade 3: Lower airway disease, or; Upper airway involvement
  * Grade 4: Lower or upper airway condition, or; Cardiovascular system involvement
  * Grade 5: Death
Number of Adverse Reactions to any medication | 12 months
  Number of Adverse Reactions to any medication administered for the treatment of AE

CONTACTS AND LOCATIONS:
Overall Officials: Ana Isabel Tabar Purroy, MD; PhD, Principal Investigator — Complejo Hospitalario de Navarra
Locations (13):
- Spain (13):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Santa Bárbara, Puertollano, Ciudad Real
  - Hospital el Bierzo, Ponferrada, León
  - Hospital Universitario de Navarra, Pamplona, Navarre
  - Hospital Universitario A Coruña, A Coruña
  - Centro Médico ASISA Dr. Lobatón, Cadiz
  - C.P.E. Virgen de la Cinta - Hospital Universitario Juan Ramón Jiménez, Huelva
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Quirón Salud Málaga, Málaga
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario de Álava, Vitoria-Gasteiz, Álava

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Subiza J, Feliu A, Subiza JL, Uhlig J, Fernandez-Caldas E. Cluster immunotherapy with a glutaraldehyde-modified mixture of grasses results in an improvement in specific nasal provocation tests in less than 2.5 months of treatment. Clin Exp Allergy. 2008 Jun;38(6):987-94. doi: 10.1111/j.1365-2222.2008.02995.x. Epub 2008 Apr 25. PMID 18445082
- [Background] Klimek L, Uhlig J, Mosges R, Rettig K, Pfaar O. A high polymerized grass pollen extract is efficacious and safe in a randomized double-blind, placebo-controlled study using a novel up-dosing cluster-protocol. Allergy. 2014 Dec;69(12):1629-38. doi: 10.1111/all.12513. Epub 2014 Oct 6. PMID 25130503
- [Background] Guzman-Fulgencio M, Caballero R, Lara B, Mena M, Tejera M, Sastre A, Subiza JL, Fernandez-Caldas E, Casanovas M. Safety of immunotherapy with glutaraldehyde modified allergen extracts in children and adults. Allergol Immunopathol (Madr). 2017 Mar-Apr;45(2):198-207. doi: 10.1016/j.aller.2016.08.008. Epub 2016 Dec 7. PMID 27939406